CLINICAL TRIAL: NCT05642897
Title: Mind Programme for Women With Breast Cancer: A Randomized Controlled Trial Testing the Programme´s Cost-effectiveness and Efficacy in Changing Psychological and Biological Outcomes
Brief Title: Mind Programme for Women With Breast Cancer
Acronym: MIND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: IPATIMUP - Instituto De Patologia E Imunologia Molecular Da Universidade Do Porto (Other)
Responsible Party: Principal Investigator, Inês A Trindade, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CINEICC-3-IAT
Record Dates: First submitted 2022-11-17; First posted 2022-12-08 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer Female
Keywords: Mindfulness; Compassion Focused Therapy; Acceptance and Commitment Therapy; biological markers; cost-effectiveness; mental health
MeSH Terms: conditions — Psychological Well-Being | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind (Experimental): The Mind programme is an ACT, mindfulness and compassion intervention for women with breast cancer. It will include 8 weekly group sessions, with the duration of 120 minutes each, and will be delivered at the Radiotherapy Service of the CHUC or through an online platform. All participants will continue on receiving the recommended medical treatment for their clinical diagnosis.
  Interventions: Behavioral: Mind
- Support group (Active Comparator): A support group intervention, with 8 weekly 90-120-minute sessions, will be delivered to the active control group at the Radiotherapy Service of the CHUC or through an online platform. All participants will continue on receiving the recommended medical treatment for their clinical diagnosis.
  Interventions: Behavioral: Support Group

INTERVENTIONS:
Behavioral: Mind — ACT, mindfulness, and compassion-based intervention
  Arms: Mind
Behavioral: Support Group — This intervention promotes the sharing of cancer-related experiences, active listening and a sense of community between participants.
  Arms: Support group

SUMMARY:
The Mind programme for cancer patients was developed by this project PI through the integration of ACT, mindfulness and CFT components specifically adapted to the needs of a cancer population. This intervention aims at improving well-being, preventing subsequent distress, and promoting adaptation to the disease and posttreatment period. A recent pilot study presented preliminary findings on this intervention, suggesting high acceptability and efficacy in improving self-reported psychological health in breast cancer patients undergoing Radiotherapy treatment. Nevertheless, this study's small sample size, methodology (inactive control group), and exclusive reliance on self-reported data limit the interpretation and generalization of results, creating an avenue for the optimization and further testing of the programme through more robust and reliable methods. The aim of this project is therefore to optimize the Mind programme taking into consideration the results from its pilot study and to conduct a Randomized Controlled Trial on the efficacy of the intervention in improving not only mental health outcomes but also biological markers, as well as on its cost-effectiveness, in women with breast cancer. The superiority of the Mind programme will be compared to a support group intervention through the analysis of changes in cancer-specific quality of life, depressive symptoms and anxiety severity, psychological experiences, and immunological and epigenetics markers related to mental health and breast cancer prognosis. All participants will receive the intervention that shows better results.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18-70;
2. primary diagnosis of BC (stages between I and III);
3. undergoing radiotherapy treatment at CHUC;
4. able to understand and answer to self-report questionnaires in Portuguese.

Exclusion Criteria:

1. currently undergoing any form of psychological intervention;
2. current diagnosis of severe psychiatric illness (psychotic disorder, bipolar disorder, substance abuse, and personality disorder) or suicidal ideation;
3. diagnosis of neurological disease.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Cancer-specific quality of life | Baseline, post-treatment (2 months after baseline), and 6-months follow-up
  EORTC QLQ-C30 - Quality of Life, the higher the score, the higher the QoL level

SECONDARY OUTCOMES:
Psychological flexibility | Baseline, post-treatment (2 months after baseline), and 6-months follow-up
  Comprehensive Assessment of Acceptance and Commitment Therapy's Processes, the higher the score, the higher psychological flexibility level
Self-compassion and mindfulness | Baseline, post-treatment (2 months after baseline), and 6-months follow-up
  Self-compassion Scale, the higher the score, the higher the self-compassion or mindfulness level
Immunological and epigenetic markers | Baseline, post-treatment (2 months after baseline) and 6-months follow-up
  Immunology indicators. Inflammatory biomarkers formerly associated with depression and anxiety (e.g., CRP, IL-6 and TNFalpha); biomarkers of the development of effective immune surveillance (e.g., IFNgamma, IL-12/18, GM-CSF); suppressive cytokines that may block the development of effective anti-tumour immune responses (e.g., IL-10, IL-4/13).
  Epigenetics indicators. Expression of miRs associated with stress response, inflammation, or BC prognosis (miR-21, miR-146a, miR-155, and miR-Let7).
General quality of life | Baseline, post-treatment (2 months after baseline), and 6-months follow-up
  EQ-5D-5L, the higher the score, the higher the QoL level
Major life events questionnaire - controlling variable | 6-months follow-up
  Major Life Event Questionnaire, the higher the score, the higher the number of major life events in the previous year
ACT processes (Hexa(in)Flex Interview) | Baseline
  Hexa(in)Flex Interview is a semi-structured interview that aims to assess qualitatively the subjective experience of the 6 core processes of the Psychological (In)Flexibility Model underlying ACT in women with breast cancer. The interview has two parts: 1) an introduction to the aims of the interview, as well as introductory questions regarding diagnostic information (e.g., duration of diagnosis, treatment phase, support network) and general coping and adaptation to the cancer diagnosis; 2) Five sections of open questions aiming to assess: experiential avoidance versus acceptance, cognitive fusion versus defusion, conceptual versus contextual self, Past and future conceptualized (auto-pilot) versus contact with present moment, and lack of values clarity and action versus commitment to valued action. Each section has instructions on how the interviewer should conduct the questioning, as well as additional tips and caveats that should be considered.
Consumption of resources and costs | Baseline, post-treatment (2 months after baseline), and 6-months follow-up
  To collect data regarding resources used by participants outside the hospital setting, the research team developed a questionnaire adapted from the UK Cancer Costs Questionnaire (UKCC) Version 2.0 (http://blogs.ed.ac.uk/ukcc). Hospital costs will be taken from clinical registries.
Depressive symptoms and anxiety severity | Baseline, post-treatment (2 months after baseline), and 6-months follow-up
  HADS, the higher the score, the higher anxiety and depression level

CONTACTS AND LOCATIONS:
Locations (1):
- Radiotherapy Service of the Coimbra University Hospital (CHUC), Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trindade IA, Soares A, Skvarc D, Carreiras D, Pereira J, Lourenco O, Sampaio F, de Sousa B, Martins TC, Boaventura P, Marta-Simoes J; Mind Project Team; Moreira H. Efficacy and cost-effectiveness of an ACT and compassion-based intervention for women with breast cancer: study protocol of two randomised controlled trials 1. Trials. 2025 Jan 3;26(1):5. doi: 10.1186/s13063-024-08626-4. PMID 39754194